CLINICAL TRIAL: NCT00849485
Title: Randomized, Open-Label, 2-Way Crossover, Bioequivalence Study of Levetiracetam 750 mg Tablet and Keppra® (Reference) Following a 750 mg Dose in Healthy Subjects Under Fed Conditions
Brief Title: Levetiracetam 750 mg Tablets Under Non-Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 50277
Record Dates: First submitted 2009-02-20; First posted 2009-02-24 (Estimated); Results first posted 2009-08-04 (Estimated); Last update posted 2009-09-11 (Estimated); Status verified 2009-09

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levetiracetam (Experimental): Levetiracetam 750 mg Tablet (test) dosed in first period followed by Keppra® 750 mg Tablet (reference) dosed in second period
  Interventions: Drug: Levetiracetam
- Keppra® (Active Comparator): Keppra® 750 mg Tablet (reference) dosed in first period followed by Levetiracetam 750 mg Tablet (test) dosed in second period
  Interventions: Drug: Keppra®

INTERVENTIONS:
Drug: Levetiracetam — 750 mg Tablet
  Arms: Levetiracetam
Drug: Keppra® — 750 mg Tablet
  Arms: Keppra®

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of a test formulation of Levetiracetam tablets versus the reference Keppra® administered as a 1 x 750 mg tablet under fed conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria

* Male or Female, smoker or non-smoker, between the ages of 18 years and 55 years.
* BMI greater than or equal to 19.0 and less than 30.0 kg/m2.

Exclusion Criteria

Subjects to whom any of the following applies will be excluded from the study:

* Clinically significant illnesses or surgery within 4 weeks of the administration of study medication.
* Any clinically significant abnormality or abnormal laboratory test results found during medical screening.
* Any reason which, in the opinion of the medical subinvestigator, would prevent the subject from participating in the study.
* Positive testing for hepatitis B, hepatitis C or HIV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, or diastolic blood pressure lower than 50 or over 90; or heart rate less than 50 bpm or over 100 bpm) at screening.
* History of significant alcohol abuse or drug abuse within one year prior to the screening visit.
* Regular use of alcohol within six months prior to the screening visit (more than fourteen units of alcohol per week [1 Unit = 150 mL of wine, 360 mL of beer or 45 mL of 40% alcohol]), or positive alcohol breath test at screening.
* Use of soft drugs (such as marijuana) within 3 months of the screening visit or hard drugs (such as cocaine, phencyclidine (PCP) and crack) within 1 year of the screening visit or positive urine drug screen at screening.
* History of allergic reactions to heparin, levetiracetam, or other related drugs.
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; examples of inhibitors: antidepressants, cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fluoroquinolones, antihistamines) within 30 days prior to the administration of the study medication.
* Use of an investigational drug or participation in an investigational study within 30 days prior to dosing.
* Clinically significant history or presence of any gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism or excretion of the drug.
* Any clinically significant history or presence of neurological, endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric or metabolic disease.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products) including natural food supplements, vitamins, garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Difficulty to swallow study medication.
* Smoking more than 25 cigarettes per day.
* Any food allergy, intolerance, restriction, or special diet, that, in the opinion of the Medical Sub-Investigator could contraindicate the subject's participation in this study.
* A depot injection or an implant of an drug within 6 months prior to administration of study medication.
* Donation of plasma (500 mL) within 30 days prior to drug administration. Donation or loss of whole blood (excluding the volume of blood that will be drawn during the screening procedures of this study) prior to administration of the study medication as follows:
* 50 mL to 500 mL of whole blood within 30 days
* more than 500 mL of whole blood within 56 days.+
* Difficulty fasting or consuming the standard meals.
* Intolerance to venipunctures.
* Clinically significant history of renal, hepatic, or cardiovascular disease, tuberculosis, epilepsy, asthma, diabetes, psychosis or glaucoma will not be eligible for this study.
* Positive urine pregnancy test at screening.
* Breast feeding subjects.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2005-11; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Audet, MD, Principal Investigator — SFBC Anapharm
Locations (1):
- SFBC Anapharm, Sainte-Foy, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Levetiracetam (Test) First: Levetiracetam 750 mg Tablet (test) dosed in first period followed by Keppra® 750 mg Tablet (reference) dosed in second period
- Keppra® (Reference) First: Keppra® 750 mg Tablet (reference) dosed in first period followed by Levetiracetam 750 mg Tablet (test) dosed in second period
Period: First Intervention
Arm/Group | Levetiracetam (Test) First | Keppra® (Reference) First
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Washout: 7 Days
Arm/Group | Levetiracetam (Test) First | Keppra® (Reference) First
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Levetiracetam (Test) First | Keppra® (Reference) First
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levetiracetam (Test) First | Keppra® (Reference) First | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 6 | 5 | 11
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 11 | 11 | 22
Region of Enrollment [Number; unit: participants]
  Canada | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: mcg/mL
Groups:
- Levetiracetam: Levetiracetam 750 mg Tablet (test) dosed in either period
- Keppra®: Keppra® 750 mg Tablet (reference) dosed in either period
Arm/Group | Levetiracetam | Keppra®
Number analyzed (Participants) | 22 | 22
mcg/mL | 19.635 (3.854) | 20.054 (4.125)
Statistical Analysis 1: Comparison: Levetiracetam vs Keppra®; Test type: Non-Inferiority or Equivalence — Using GLM procedures in SAS, analysis of variance (ANOVA)was performed on log-transformed AUC0-t, AUC0-inf and Cmax at the significance level of 0.05; Geometric Test/Ref Ratio x 100 = 98.0, 90% CI [94.5 to 102] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | Levetiracetam | Keppra®
Number analyzed (Participants) | 22 | 22
mcg*h/mL | 186.758 (30.682) | 186.899 (31.029)
Statistical Analysis 1: Comparison: Levetiracetam vs Keppra®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Test/Ref Ratio x 100 = 99.9, 90% CI [97.6 to 102] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | Levetiracetam | Keppra®
Number analyzed (Participants) | 22 | 22
mcg*h/mL | 176.267 (31.911) | 174.729 (33.259)
Statistical Analysis 1: Comparison: Levetiracetam vs Keppra®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Test/Ref Ratio x 100 = 101, 90% CI [98.1 to 104] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.